CLINICAL TRIAL: NCT00466713
Title: Defining the Role of Insulin Resistance in 'Idiopathic' Dilated Cardiomyopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: concern over safety of rosiglitazone in heart failure
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael Fowler, Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 5367
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Dilated Cardiomyopathy
Keywords: Nonischemic dilated cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rosiglitazone therapy

SUMMARY:
This study will investigate the effects of rosiglitazone, a medicine commonly used to treat type 2 diabetes, on the utilization of glucose by the heart in patients with heart failure which is not due to heart attacks. The primary purpose of the study is to determine whether treatment with an insulin-sensitizing medication will improve the heart's ability to metabolize glucose (sugar).

DETAILED DESCRIPTION:
Nondiabetic patients with nonischemic cardiomyopathy who are insulin-resistance or insulin-sensitive based on a fasting homeostasis model assessment (HOMA) value are eligible for the trial. At baseline, a 6-minute walk test is performed, followed by assessment of coronary flow reserve with ammonia-PET imaging before/after adenosine infusion. Subjects are then given an oral glucose load (75g), followed by PET imaging with F-18-fluoro-2-deoxyglucose (FDG). Subjects then begin taking rosiglitazone 4 mg qd x 12 weeks, after which the 6-minute walk test & PET imaging is repeated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nonischemic dilated cardiomyopathy, current NYHA class I-II congestive heart failure
* History of Stage C-D heart failure with EF ≤ 40% during the course of the disease
* Treatment with a stable comprehensive heart failure regimen for at least 3 months (including beta-blockers and ACE-inhibitors or angiotensin receptor blockers unless intolerant)
* Age > 18 yrs

Exclusion Criteria:

* Cardiomyopathy due to one of the following:

  * Ischemic heart disease
  * Primary valvular lesion
  * Hypertrophic cardiomyopathy
* Cardiac resynchronization within the last 3 months
* Transaminase values > 2.5 x upper limit of normal or history of liver disease
* Diagnosis of diabetes mellitus by:

  * Diabetes previously diagnosed per patient history
  * 2 or more fasting glucose values > 125 mg/dl
* Current NYHA class III or IV heart failure
* Serum creatinine > 1.6 mg/dl
* History of heart transplantation
* Pregnancy or active breast feeding
* Hospitalization for decompensated heart failure within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Myocardial glucose uptake (intrasubject before/after rosiglitazone)
Myocardial glucose uptake (between insulin-resistant & insulin-sensitive groups)

SECONDARY OUTCOMES:
Coronary flow-reserve
6-minute walk time

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fowler, MB, Principal Investigator — Stanford University
Locations (1):
- Stanford University Hospital, Stanford, California, United States